CLINICAL TRIAL: NCT02345330
Title: A Multicenter Phase II Trial of Intratumoral pIL-12 Electroporation in Treatment-Refractory Metastatic and Unresectable SCC of the Head and Neck
Brief Title: Trial of pIL-12 Electroporation in Squamous Cell Carcinoma of the Head and Neck (IL12HNSCC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to company resource constraints
Sponsor: OncoSec Medical Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMS-I130
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Results first posted 2018-01-03 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tavokinogene Telseplasmid (tavo) Electroporation (EP) (Experimental): Participants received tavo intratumorally followed immediately by electroporation (EP) on Days 1, 8, and 15 in a 6-week cycle for up to 9 cycles.
  Interventions: Biological: Tavokinogene Telseplasmid (tavo); Device: OncoSec Medical System (OMS)

INTERVENTIONS:
Biological: Tavokinogene Telseplasmid (tavo) — Patients received intratumoral injection(s) of tavo.
  Other Names: pIL-12; IL-12 gene; plasmid DNA encoding human interleukin-12; plasmid IL-12; interleukin-12 gene
Device: OncoSec Medical System (OMS) — Electroporation via OMS was performed immediately following intratumoral injection of tavo. A sterile applicator containing 6 stainless steel electrodes arranged in a circle were placed around the tumor. The applicator was connected to the OMS power supply and six pulses were administered to each tumor lesion at the approximate point of tavo injection.
  Other Names: MedPulser

SUMMARY:
This study will assess the safety and effectiveness of ImmunoPulse IL-12® in treatment-refractory metastatic and unresectable squamous cell carcinoma of the head and neck (HNSCC). ImmunPulseIL12® is the combination of intrtumoral interleukin-12 gene (also known as tavokinogene telseplasmid [tavo]) and in vivo electroporation-mediated plasmid deoxyribonucleic acid [DNA] vaccine therapy (tavo-EP) administered using the OncoSec Medical System (OMS). Intratumoral tavo is a gene therapy approach to directly induce a pro-inflammatory response within a tumor to initiate and/or enhance anti-tumor immunity.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological diagnosis of squamous cell carcinoma (SCC) of head and neck with American Joint Committee on Cancer (AJCC) Stage III, IVA or IVB and not amenable to surgical resection or locoregional radiation therapy with curative intent.
2. Patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
3. Patients must have at least one tumor accessible for intratumoral injection and EP on investigator's assessment.
4. Patients must have at least one additional lesion (measurable by RECIST v1.1 or non-target) identified as a control untreated lesion to be left untreated and followed for response.
5. Patients may have had prior chemotherapy or immunotherapy or radiation therapy. Any drug-related adverse events (AEs) identified during prior therapy must have been well-controlled (typically resolution to ≤ Grade 2), or resolved upon investigator review prior to initiation of the study therapy.
6. Patients must have platinum-refractory disease defined as disease progression within 12 months platinum-based chemoradiation with curative intent or any disease progression on platinum-based chemotherapy in the absence of radiation.
7. Age ≥ 18 years old.
8. Patients must have agreed to a new biopsy of tumor (deemed accessible and safe for biopsy by the investigator's assessment) and allowing acquired tissue to be used for biomarker analysis. If the biopsied lesions were previously irradiated, they must demonstrate either radiographic or pathological evidence of recurrent or residual disease.
9. No systemic antineoplastic therapy may have been received between the time of biopsy and the first administration of study treatment.
10. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
11. Life expectancy of at least 3 months.
12. Adequate organ function.
13. Female patient of childbearing potential has a negative pregnancy test within 14 days prior to the start of study drug.
14. Women of child-bearing potential and men must agree to use adequate contraception.
15. Able to give informed consent.

Exclusion Criteria:

1. Prior therapy with IL-12 or prior gene therapy.
2. Concurrent ongoing administration of systemic therapy (e.g. chemotherapy), or radiation therapy.
3. Evidence of significant active infection (e.g., pneumonia, cellulitis, wound abscess, etc.) at time of study entry.
4. Pregnant or breast-feeding women are excluded.
5. Patients with electronic pacemakers or defibrillators are excluded.
6. Significant disease or uncontrolled disease, i.e. cardiovascular renal, hepatic, endocrine, metabolic, neurologic; or other significant disease that would limit the patients ability to participate in the study as determined by the investigator or medical monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2016-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Chicago Medical Center, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 21 May 2015 to 14 November 2016.
Period: Overall Study
Arm/Group | Tavokinogene Telseplasmid (Tavo) Electroporation (EP)
Started | 4
Completed | 1
Not Completed | 3
Not completed — Death | 1
Not completed — Progressive Disease | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Arm/Group | Tavokinogene Telseplasmid (Tavo) Electroporation (EP)
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (4.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (BORR) by RECIST v1.1
Description: BORR is defined as the percentage of participants with evaluable lesions that achieved a complete response (CR) or partial response (PR) as assessed by the investigator using Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR: Disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR: At least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions.
Time Frame: Every 6 weeks until disease progression, death, withdrawal of consent or study termination (up to 14.5 months)
Population: Due to early termination of the study BORR by RECIST v1.1 data was not collected and reported.
Arm/Group | Tavokinogene Telseplasmid (Tavo) Electroporation (EP)
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, medical treatment or procedure and which did not necessarily have to have had a causal relationship with this treatment. An adverse event could have, therefore, been any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, medical treatment or procedure whether or not considered related to the medicinal product. An SAE was defined an any untoward medical occurrence that at any dosage resulted in one or more of the following: death, A life-threatening adverse event (real risk of dying), inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital anomaly, required intervention to prevent permanent impairment of damage.
Time Frame: From first study treatment to 30 days after the last study treatment (up to 14.5 months)
Population: All enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tavokinogene Telseplasmid (Tavo) Electroporation (EP)
Number analyzed (Participants) | 4
Participants
  AEs | 4
  SAEs | 1

3. Secondary Outcome: Best Overall Response Rate (BORR) by Immune-related Response Criteria (irRC)
Description: BORR is defined as the percentage of participants with evaluable lesions that achieved a complete response (CR) or partial response (PR) as assessed by the investigator using irRC criteria. CR: complete disappearance of all lesions (whether measurable or not) and the absence of new lesions for at least 4 weeks duration, confirmed by additional scan and visit 4 to 6 weeks after first documentation of CR. PR: ≥50% decrease in the product of the diameters from baseline.
Time Frame: Every 6 weeks until disease progression, death, withdrawal of consent or study termination (up to 14.5 months)
Population: Due to early termination of the study BORR by irRC data was not collected and reported.
Arm/Group | Tavokinogene Telseplasmid (Tavo) Electroporation (EP)
Number analyzed (Participants) | 0

4. Secondary Outcome: Regression Rate of Treated and Untreated Lesions
Description: The treated (injected, electroporated) lesion regression rate is defined as the percentage of patients who had at least one treated lesion that decreased in longest dimension by ≥ 30%. The untreated (non-injected, non-electroporated) lesion regression rate is defined as the percentage of patients who had at least one untreated lesion that decreased in longest dimension by ≥ 30%.
Time Frame: Every 6 weeks until disease progression, death, withdrawal of consent or study termination (up to 14.5 months)
Population: Due to early termination of the study regression rate data was not collected and reported.
Arm/Group | Tavokinogene Telseplasmid (Tavo) Electroporation (EP)
Number analyzed (Participants) | 0

5. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Progression free survival (PFS) time is defined as the duration between the date of treatment initiation (Study Day 1) to the first date of either disease progression at either local or any distant sites, or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Patients were censored at their date of last assessment, if they were alive and without evidence of disease progression.
Time Frame: From start of study treatment weeks until disease progression, death, withdrawal of consent or study termination (up to 14.5 months)
Population: Due to early termination of the study PFS data was not collected and reported.
Arm/Group | Tavokinogene Telseplasmid (Tavo) Electroporation (EP)
Number analyzed (Participants) | 0

6. Secondary Outcome: Median Time to Progression (TTP)
Description: TTP is defined as the number of days between the treatment initiation date (Study Day 1) and the earliest date of documented disease progression as defined by RECIST 1.1 or death that is not associated with prior disease progression. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: as for outcome 5
Population: Due to early termination of the study TTP data was not collected and reported.
Arm/Group | Tavokinogene Telseplasmid (Tavo) Electroporation (EP)
Number analyzed (Participants) | 0

7. Secondary Outcome: Median Overall Survival (OS)
Description: Overall survival is defined as the time in days from the date of first study drug administration to the date of death.
Time Frame: From the start of study treatment until death
Population: Due to early termination of the study overall survival data was not collected and reported.
Arm/Group | Tavokinogene Telseplasmid (Tavo) Electroporation (EP)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first study treatment to 30 days after the last study treatment (up to 14.5 months)
Arm/Group | Tavokinogene Telseplasmid (Tavo) Electroporation (EP)
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tavokinogene Telseplasmid (Tavo) Electroporation (EP) (N=4)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tavokinogene Telseplasmid (Tavo) Electroporation (EP) (N=4)
Nausea (Gastrointestinal disorders) | 1
Injection site bruising (General disorders) | 1
Injection site haemorrhage (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Procedural pain (Injury, poisoning and procedural complications) | 2
Paraesthesia (Nervous system disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less